CLINICAL TRIAL: NCT06953336
Title: Improving Dietary Quality and Health Outcomes: A Fruit and Vegetable Voucher Program for Kidney Transplant Patients With Food Insecurity.
Brief Title: Vouchers for Improving Transplant Access to Lifestyle Nutrition - Kidney Transplant
Acronym: VITAL-KT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-43473; P0580734 (Other Grant/Funding Number: Agency of Healthcare Research and Quality)
Record Dates: First submitted 2025-04-21; First posted 2025-05-01 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Food Insecurity; Kidney Transplant
Keywords: Food Vouchers; Food Insecurity; Kidney Transplant; Dietary Quality; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Fruit

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Food Voucher Intervention Arm (Experimental): Participants in this arm will receive monthly food vouchers in the form of an Electronic Benefit Transfer (EBT) card, which will be mailed to their home and refilled each month for a total of 6 months. The EBT cards are provided and managed by an external community-based organization in partnership with the research team. The voucher amount is intended to supplement household food purchases and reduce food insecurity. The intervention targets pediatric and young adult kidney transplant recipients who have screened positive for food insecurity within the past 6 months. The participants will use the vouchers, and both pre- and post-intervention surveys will be administered to assess food security status and dietary quality. This supportive care intervention is designed to enhance nutritional support and promote stability during the post-transplant period.
  Interventions: Other: Fruit and Vegetable Voucher Support Program

INTERVENTIONS:
Other: Fruit and Vegetable Voucher Support Program — Participants will receive a monthly food voucher in the form of an Electronic Benefit Transfer (EBT) card, mailed to their home and refilled each month for 6 months. The EBT cards are provided and managed by an external community-based organization in partnership with the research team. The intervention is designed to supplement household food purchases, reduce food insecurity, and support nutritional well-being among pediatric and young adult kidney transplant recipients who have recently screened positive for food insecurity. Pre- and post-intervention surveys will be used to assess food security status and dietary quality.

SUMMARY:
This study evaluates the effect of a six-month fruit and vegetable voucher program on satisfaction, dietary quality, and health outcomes among pediatric and young adult kidney transplant recipients experiencing food insecurity.

DETAILED DESCRIPTION:
This is a single-arm, prospective interventional study enrolling 18 participants aged 6 to 25 years who have undergone kidney transplantation and screened positive for food insecurity within the past six months.

Participants will receive monthly fruit and vegetable vouchers for six months, distributed via Electronic Benefit Transfer (EBT) cards. The EBT cards, managed by an external partner, will be automatically reloaded monthly and be redeemable at participating retailers.

Data collection will include participant-reported satisfaction surveys post-intervention, food security and dietary quality assessments at baseline and study end, biophysical outcomes (BMI, blood pressure) from routine clinical care, laboratory markers related to kidney and nutritional health (serum potassium, phosphorus, magnesium, albumin, bicarbonate, fasting glucose or HbA1c, and creatinine/GFR), tacrolimus variability to serve as a proxy for medication adherence.

No extra clinical visits or lab draws beyond standard care are required. The findings aim to inform future strategies to address food insecurity in transplant populations.

ELIGIBILITY:
Inclusion Criteria:

* Age: Children and young adults aged 2 to 25 years who have received a kidney transplant.
* Food Insecurity: Patients who have screened positive for food insecurity (FI) within the past six months, based on the Hunger Vital Sign
* Patients who are currently receiving care at the transplant center and whose caregivers (if the patient is less than 18 years of age) are willing to participate in the intervention.
* Caregivers of non-adult patients

Exclusion Criteria:

* Patient being on a diet consisting of only total parenteral nutrition or tube feeds.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction Difference | From enrollment to the end of treatment at 6 months
  Participant satisfaction with the food voucher program assessed through a survey administered by the end of the 6-month intervention period. This survey will evaluate participants' overall satisfaction with the EBT card, including the perceived impact on food security, ease of use, and the perceived value of the program.

SECONDARY OUTCOMES:
Number of participants who screen positively for food insecurity | From enrollment to the end of treatment at 6 months
  Food security status will be assessed using a validated food security questionnaire at baseline and post-intervention. This measure will capture changes in household food access and adequacy as a result of the intervention.
Dietary Quality Difference | From enrollment to the end of treatment at 6 months
  Dietary quality will be assessed using self-reported dietary intake questions included in the pre- and post-intervention surveys. This measure will provide insight into any changes in the participants' food choices and nutritional habits due to the intervention, focusing on the amount of monthly fruit and vegetable intake.
Number of participants who screen positively for nutrition insecurity | From enrollment to the end of treatment at 6 months
  Nutrition security status will be assessed using validated nutrition security questions within the pre- and post-surveys.
Body mass index (BMI) Difference | At baseline and 6 months.
  Weight and height will be combined to report BMI in kg/m^2.
Blood pressure difference | From enrollment to the end of treatment at 6 months
  Difference of systolic and diastolic blood pressure as measured in mmHg.

OTHER OUTCOMES:
Serum Creatinine and GFR difference | From enrollment to the end of treatment at 6 months
  Kidney function assessed through serum creatinine and estimated GFR.
Tacrolimus Variability (Proxy for Medication Adherence) | From enrollment to the end of treatment at 6 months
  Tacrolimus variability will be assessed by measuring fluctuations in tacrolimus blood levels during the study period. Variability in tacrolimus levels can serve as a proxy for medication adherence in pediatric kidney transplant recipients. Stable tacrolimus levels typically reflect better adherence to prescribed medication regimens, and variability can indicate missed doses or inconsistent adherence.
HbA1c difference | From enrollment to the end of treatment at 6 months
  Glycemic control assessed by difference of HbA1c percent (%) values
Serum potassium difference | From enrollment to the end of treatment at 6 months
  Difference on serum potassium as measured in mEq/L
Serum magnesium difference | From enrollment to the end of treatment at 6 months
  Serum magnesium difference as measured in mg/dL.
Serum bicarbonate difference | From enrollment to the end of treatment at 6 months
  Serum bicarbonate difference measured in CO2 content in blood in mEq/L
Changes in medications | From enrollment to the end of treatment at 6 months
  Changes in medications such as blood rpessure mendications and supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Eva Glenn Lecea, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stein R, Finnie RKC, Harmon S, Peng Y, Pritchard C, Vecsey H, Emmons KM, Hargarten S, Simon MA, Blanck HM, Harris DM, Bellows L, Coleman-Jensen A, Fleischhacker S, Koenings MM, Odoms-Young A, Seligman HK, Grant C, Powell A; Community Preventive Services Task Force. Impact of Fruit and Vegetable Incentive Programs on Food Insecurity, Fruit and Vegetable Consumption, and Health Outcomes: A Community Guide Systematic Review. Am J Prev Med. 2025 Mar;68(3):627-637. doi: 10.1016/j.amepre.2024.11.016. Epub 2024 Dec 2. PMID 39631447
- [Background] Twichell S, Hunt EAK, Ciurea R, Somers MJG; NAPRTCS investigators. Rapid Weight Gain After Pediatric Kidney Transplant and Development of Cardiometabolic Risk Factors Among Children Enrolled in the North American Pediatric Renal Trials and Collaborative Studies Cohort. Pediatr Transplant. 2025 Feb;29(1):e70005. doi: 10.1111/petr.70005. PMID 39729540
- [Background] Ridberg RA, Levi R, Marpadga S, Akers M, Tancredi DJ, Seligman HK. Additional Fruit and Vegetable Vouchers for Pregnant WIC Clients: An Equity-Focused Strategy to Improve Food Security and Diet Quality. Nutrients. 2022 Jun 1;14(11):2328. doi: 10.3390/nu14112328. PMID 35684128
- [Background] Basu S, Akers M, Berkowitz SA, Josey K, Schillinger D, Seligman H. Comparison of Fruit and Vegetable Intake Among Urban Low-Income US Adults Receiving a Produce Voucher in 2 Cities. JAMA Netw Open. 2021 Mar 1;4(3):e211757. doi: 10.1001/jamanetworkopen.2021.1757. PMID 33749765